CLINICAL TRIAL: NCT00794079
Title: Omega-3 Fatty Acids and Muscle Protein Synthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Longer Life Foundation (Other); American Federation for Aging Research (Other); Reliant Pharmaceuticals (Industry)
Responsible Party: Bettina Mittendorfer, PhD, WashingtonU
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 06-1147
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-08

CONDITIONS: Healthy
Keywords: Healthy volunteers; young adults; Aged
MeSH Terms: interventions — Fatty Acids, Omega-3; Omacor; Corn Oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): omega-3 fatty acids
  Interventions: Dietary Supplement: omega-3 fatty acids
- B (Placebo Comparator): corn oil
  Interventions: Dietary Supplement: corn oil

INTERVENTIONS:
Dietary Supplement: omega-3 fatty acids — 4 grams per day for 8 weeks
  Other Names: Lovaza
  Arms: A
Dietary Supplement: corn oil — 4 grams per day for 8 weeks
  Arms: B

SUMMARY:
The purpose of this study is to determine whether omega-3 fatty acid supplementation influences muscle protein synthesis rates in young and older adults.

DETAILED DESCRIPTION:
Loss of muscle mass is a normal consequence of aging. The decline in muscle mass is estimated to be 0.2-0.5% per year from 60 years old onwards in healthy subjects with the decline worsened by chronic illness, poor appetite and diet, and reduced physical activity in the elderly. Increased morbidity is demonstrable with as little as a 5% loss of muscle mass - therefore, treatments that can prevent or slow the progression of muscle loss with aging are much desired.

A major cause for loss of muscle mass in advanced age appears to be an impaired ability to stimulate the synthesis of muscle protein in response to increased levels of amino acids (the building blocks of proteins) and insulin as occurs after eating because of low-grade inflammation and insulin resistance in muscle of old persons. We propose that long-chain omega-3 polyunsaturated fatty acids (fish oil) slow the loss of muscle mass because fish oil has anti-inflammatory properties and increases the sensitivity of muscle protein synthesis to insulin and amino acids. We will test this by studying the effect of fish oil supplementation on the muscle protein synthesis process in young and older adults.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) < 30 kg/m2;
* Age 18-45 yr; or
* Age 65-85 yr

Exclusion Criteria:

* Those taking medications known to affect substrate metabolism or medications that may confound the findings from our study (synthetic steroids, glucocorticoids etc.);
* Those with evidence of significant organ system dysfunction (e.g. diabetes mellitis, cirrhosis, hypo- or hyperthyroidism; hypertension);
* Body mass index > 30 kg/m2
* Age <18 yr, 45-65 yr or > 85 yr
* Those performing >1.5h of exercise/wk

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of omega-3 fatty acid supplementation on skeletal muscle protein synthesis rates both in the basal, postabsorptive state and in response to infusion of insulin and amino acids in young and older adults | Measurements taken prior to and following 8 weeks of supplementation

SECONDARY OUTCOMES:
Evaluate the effect of omega-3 fatty acid supplementation on anabolic signaling pathways in skeletal muscle | Measurements taken prior to and following 8 weeks of supplementation
Evaluate the effect of omega-3 fatty acid supplementation on inflammatory cytokines in the systemic circulation and inflammatory signaling pathways in skeletal muscle | Measurements taken prior to and following 8 weeks of supplementation
Compare muscle protein synthesis rates between men and women in the basal, postabsorptive state and in response to insulin and amino acid infusion | prior to supplementation only

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Mittendorfer, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in Saint Louis, St Louis, Missouri, United States

REFERENCES:
- [Result] Smith GI, Atherton P, Reeds DN, Mohammed BS, Rankin D, Rennie MJ, Mittendorfer B. Dietary omega-3 fatty acid supplementation increases the rate of muscle protein synthesis in older adults: a randomized controlled trial. Am J Clin Nutr. 2011 Feb;93(2):402-12. doi: 10.3945/ajcn.110.005611. Epub 2010 Dec 15. PMID 21159787
- [Result] Smith GI, Atherton P, Reeds DN, Mohammed BS, Rankin D, Rennie MJ, Mittendorfer B. Omega-3 polyunsaturated fatty acids augment the muscle protein anabolic response to hyperinsulinaemia-hyperaminoacidaemia in healthy young and middle-aged men and women. Clin Sci (Lond). 2011 Sep;121(6):267-78. doi: 10.1042/CS20100597. PMID 21501117
- [Result] Smith GI, Atherton P, Reeds DN, Mohammed BS, Jaffery H, Rankin D, Rennie MJ, Mittendorfer B. No major sex differences in muscle protein synthesis rates in the postabsorptive state and during hyperinsulinemia-hyperaminoacidemia in middle-aged adults. J Appl Physiol (1985). 2009 Oct;107(4):1308-15. doi: 10.1152/japplphysiol.00348.2009. Epub 2009 Jul 30. PMID 19644030